CLINICAL TRIAL: NCT00509665
Title: A Phase II Study of Gemcitabine in Combination With Doxorubicin for Patients With Head and Neck Cancer
Brief Title: Gemcitabine and Doxorubicin in Treating Patients With Recurrent or Progressive Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000558049; MUSC-100838
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine+doxorubicin (Experimental)
  Interventions: Drug: doxorubicin hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: doxorubicin hydrochloride — given as 25mgm2 IV on days 1 and 8 of each 21-day cycle.
Drug: gemcitabine hydrochloride — given as 100mg/m2 IV over days 1 and 8 of each 21 day cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with doxorubicin works in treating patients with recurrent or progressive head and neck cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed head and neck cancer

  * Recurrent or progressive disease
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* Must have received prior platinum-based chemotherapy regimen (cisplatin or carboplatin) with or without radiotherapy, unless the patient was deemed unsuitable for platinum-based therapy due to renal dysfunction or other clinical contraindication

Exclusion criteria:

* Known brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status (PS) ≤ 2 OR Karnofsky PS ≥ 60%
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/µL
* Total bilirubin ≤ 1.5 mg/dL
* AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal
* Creatinine ≤ 2 mg/dL OR creatinine clearance ≥ 30 mL/min
* Females of reproductive potential must not plan on conceiving children during study treatment period and must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of the study

Exclusion criteria:

* Not pregnant or breastfeeding
* History of allergic reaction attributed to compounds of similar chemical or biological composition to gemcitabine hydrochloride or doxorubicin hydrochloride
* Lower than normal cardiac ejection fraction

  * Patients must have an echocardiogram or MUGA scan prior to the use of study drugs
* Uncontrolled intercurrent illness that would limit compliance with study requirements including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation
* Clinical AIDS or known positive HIV serology

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Recovered from prior therapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 30 days since prior experimental agents
* At least 4 weeks since prior radiotherapy for palliation or for the primary tumor

Exclusion criteria:

* Prior gemcitabine hydrochloride or doxorubicin hydrochloride
* Concurrent hormones or other chemotherapeutic agents, except for steroids given for adrenal failure, hormones given for non-disease-related conditions (e.g., insulin for diabetes), or intermittent use of dexamethasone as an antiemetic
* Concurrent palliative radiotherapy
* Other concurrent investigational or commercial agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Brien, Principal Investigator — Medical University of South Carolina
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Saddoughi SA, Garrett-Mayer E, Chaudhary U, O'Brien PE, Afrin LB, Day TA, Gillespie MB, Sharma AK, Wilhoit CS, Bostick R, Senkal CE, Hannun YA, Bielawski J, Simon GR, Shirai K, Ogretmen B. Results of a phase II trial of gemcitabine plus doxorubicin in patients with recurrent head and neck cancers: serum C(1)(8)-ceramide as a novel biomarker for monitoring response. Clin Cancer Res. 2011 Sep 15;17(18):6097-105. doi: 10.1158/1078-0432.CCR-11-0930. Epub 2011 Jul 26. PMID 21791630

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine+Doxorubicin
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 57 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria in Solid Tumors (RECIST) for target lesions assessed by CT or MRI: Complete Response (CR) is the disappearance of all target lesions (TL) and non-target lesions (NTL); Partial Response (PR) is defined by either a CR of TL and stable disease (SD) in NTL or PR of TL and non-progressive disease (PD) in NTL. Response rate is the sum of CR + PR as defined above.
Time Frame: Every 6 weeks from the time of initial treatment for up to 8 months
Population: patients who were on study at the time of response assessment
Measure: Number; unit: participants
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 17
participants | 4

2. Secondary Outcome: Duration of Response
Time Frame: Every 6 weeks for up to 8 months
Population: data for this endpoint was not collected
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Time Frame: Through the end of follow up, for an average of 8 months
Population: Only patients who had re-staging scans are included in the number of participants analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 17
months | 1.6 [1.4 to 4.2]

4. Secondary Outcome: Overall Survival
Time Frame: From the time of initial therapy until the time of death.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 18
Months | 5.6 [3.8 to 18.2]

5. Secondary Outcome: Number of Patients Who Had Greater Than Grade 2 Toxicity
Time Frame: from time of initial treatment until end of study, an average of 6 months
Population: Patients who were treated on study and had greater than grade 2 toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 18
Participants | 10

6. Secondary Outcome: Correlation of Cytoxocity With Cell-cycle Arrest
Time Frame: prior to first dose of drug and every 6 weeks up to 6 months
Population: data for this endpoint was not collected
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 0

7. Secondary Outcome: Correlation of Cytotoxicity With Apoptosis in Cancer Cells
Time Frame: prior to first dose of drug and every 6 weeks for up to 6 months
Population: Data for this endpoint was not collected
Arm/Group | Gemcitabine+Doxorubicin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Prior to each cycle while on treatment for an average of 6 months
Arm/Group | Gemcitabine+Doxorubicin
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine+Doxorubicin (N=18)
neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine+Doxorubicin (N=18)
fatigue (General disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 4 (4)
leukopenia (Blood and lymphatic system disorders) | 3 (3)
anemia (Blood and lymphatic system disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 1 (1)
vomitting (Gastrointestinal disorders) | 1 (1)
infection (Infections and infestations) | 2 (2)
DVT (Vascular disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes